CLINICAL TRIAL: NCT05992311
Title: Clinical Evaluation of Montelukast on Cognitive and Mood Dysfunction and Neuroinflammation in Veterans With Gulf War Illness (GWI)
Brief Title: Clinical Evaluation of Montelukast in Veterans With Gulf War Illness
Acronym: (GWI)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Texas A&M University (Other)
Responsible Party: Principal Investigator, Drew Helmer, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-51973; CDMRP-GW210062 (Other: Congressionally Directed Medical Research Program)
Record Dates: First submitted 2023-07-28; First posted 2023-08-15 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Gulf War Syndrome
Keywords: Montelukast
MeSH Terms: conditions — Persian Gulf Syndrome | interventions — montelukast

STUDY DESIGN:
Intervention Model Description: Double blind, placebo-controlled, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study group assignment will be determined by the research pharmacist using a random number generator within blocks of four participants. Participant group assignment will be disclosed only at time of data analysis or in case of emergency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Montelukast Group (Experimental): Montelukast two capsules of 20 mg (40 mg total) taken by mouth once daily for ten weeks
  Interventions: Drug: Montelukast
- Placebo Group (Placebo Comparator): Microcrystalline cellulose two capsules taken by mouth once daily for ten weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Montelukast — This group will receive the montelukast treatment.
  Other Names: Singulair
  Arms: Montelukast Group
Other: Placebo — This group will receive a placebo pill instead of montelukast
  Arms: Placebo Group

SUMMARY:
The study addresses the pre-clinical promise of Montelukast (MLK) for improving brain function in veterans with Gulf War Illness (GWI). MLK, a US Food and Drug administration (FDA)-approved drug for asthma, has shown efficacy in an animal model of GWI to improve cognitive and mood function through modulation of leukotriene signaling and suppression of neuroinflammation.

DETAILED DESCRIPTION:
Background: Approximately 30% of Gulf War Veterans (1990-1991) suffer from Gulf War Illness (GWI), a chronic condition characterized by disabling symptoms in multiple domains. Animal models and human data suggest a prominent neuroinflammatory basis for many of the symptoms of GWI. Preliminary data from an established GWI rat model demonstrates the involvement of increased leukotriene signaling in the brain and its potential as a marker of neuroinflammation when detected in neuron- and astrocyte-derived extracellular vesicles present in the peripheral blood. MLK, an FDA-approved drug for asthma, has shown efficacy in an animal model of GWI to improve cognitive and mood function through modulation of leukotriene signaling and suppression of neuroinflammation. MLK has a strong safety record and has been recognized for its potential as a modulator of neurodegeneration in human disease and is, therefore, a promising intervention for GWI.

Hypothesis/Objective: Examine the impact of MLK on cognition, quality of life, and symptoms of depression and anxiety in Veterans with GWI and test for changes in brain-specific leukotrienes (markers of neuroinflammation) detectable in the extracellular vesicles circulating in the peripheral blood.

Specific Aim 1: To evaluate the effect of MLK on cognitive function, functional status and mood in veterans with GWI using validated neurocognitive and self-reported measures consistent with the GWI Common Data Elements.

Specific Aim 2: To examine the antiinflammatory effects of MLK on the brain. The investigators will evaluate neuron-derived extracellular vesicles and astrocyte-derived extracellular vesicles in blood samples from Veterans with GWI receiving MLK or placebo treatment.

Study Design: 1:1 randomized, double-blind, placebo controlled trial of 80 Veterans who meet both the Kansas and Center for Disease Control (CDC) definition of GWI and report cognitive dysfunction treated with either: 1) two capsules of 20 mg of MLK or 2) two capsules of matched placebo taken daily for 10 weeks. Participants will be recruited to participate at Michael E. DeBakey VA Medical Center (MEDVAMC) in Houston, TX, using best practices including Veteran community outreach and engagement, active recruitment from local and national VA databases, and a strong social media presence. Participants will be screened for eligibility by phone and attend only two in-person evaluations (self-reported instruments, blood draw, and neuropsychology tests) with regular phone contact throughout study enrollment. Blood specimens will be obtained, and plasma processed at MEDVAMC, and shipped to Texas A&M University College of Medicine (TAMU-COM) for specialized assays. Data will be maintained, managed and analyzed by the MEDVAMC team in collaboration with the TAMU team.

Impact: The findings from the proposed research will advance the understanding of the pathophysiology, validate the use of extracellular vesicle assays as a biomarker of central nervous system inflammation, and advance a potential treatment (i.e., MLK) for a specific putative underlying mechanism of GWI. The short-term impact will be an important validation of the theory of neuroinflammation as central pathophysiology of GWI through the tested hypotheses. The longer-term impact of the proposed work includes a relatively short timeline to the use of MLK as a specific treatment for GWI. Because MLK is already FDA approved and safe, if findings from this project support the safety, tolerability, and efficacy of MLK in Veterans with GWI, a definitive randomized controlled trial confirming its efficacy would be warranted.

ELIGIBILITY:
Inclusion Criteria:

* Gulf War Veterans of the U.S. military deployed on military orders to the Persian Gulf Region between August 2, 1990, and December 31, 1991
* Diagnosed with GWI according to the CDC and modified Kansas criteria as recommended by the Institute of Medicine (IOM), that is, endorse multiple or moderate-to-severe symptoms, with symptom onset during or after deployment to the Persian Gulf region in 1990-1991, persisting for six months or longer, in at least 3 of 6 domains:

  1. fatigue/sleep disturbances
  2. neurological/cognitive/mood symptoms
  3. somatic pain
  4. gastrointestinal problems
  5. respiratory symptoms
  6. skin symptoms
* Self-reported cognitive dysfunction based on a T-score of 40 or less on the PROMIS v2.0 Cognitive Function 8a short form
* Be able to:

  * provide written consent and be able to communicate with the research team in verbal and written English
  * attend the two in-person study encounters
  * have reliable telephone service for the eight weekly telephone encounters

Exclusion Criteria:

* Diagnosed by a physician with any chronic condition that may explain their profile of symptoms or prevent their ability to accurately report them including:

  * chronic autoimmune conditions
  * systemic inflammatory conditions
  * cancer not in remission at least 5 years
  * congestive heart failure
  * anemia
  * multiple sclerosis
  * amyotrophic lateral sclerosis (ALS)
  * poorly controlled diabetes
  * post-chemo or radiation syndromes
  * sickle cell anemia
  * symptomatic Coronary Artery Disease (CAD)
  * chronic liver disease
  * chemical insufficiency
  * morbid obesity (body mass index (BMI) >= 40)
  * human immunodeficiency virus (HIV)
  * alcohol/substance use disorder/stimulant/opioid/other depressant misuse in the past year
  * major mental health condition (e.g., psychosis, suicidal ideations, major depressive disorder) that interferes with their ability to accurately report symptoms
  * hospitalized or undergoing invasive procedures in the past 12 months due to exacerbations of any chronic conditions (such as diabetes, coronary artery disease, hypertension, or emphysema)
  * elevated liver enzymes (2.5 times upper limit of normal) at baseline visit
  * estimated glomerular filtration rate less than 60 ml/min/1.73 sqm at baseline visit
  * hemoglobin less than 10 g/L at baseline visit
  * evidence of poorly controlled chronic conditions listed above, or others that may mimic GWI as per the PI, either by self-report, Veterans Health Administration (VHA) electronic health record information review, laboratory testing or physical examination
* Changes in medications for chronic conditions in the 3 months preceding enrollment (based on self-report)
* Suicidal ideation based on their responses on the Columbia Suicide Risk Inventory
* Prescribed or taking Montelukast in the past 6 months for any reason
* Taking 2 or more medications with moderate interactions with Montelukast
* Pregnancy or intention to become pregnant
* Active homicidal ideation
* COVID-19 illness (confirmed or suspected) without recovery to pre-COVID health status

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Leukotriene concentration | taken at baseline (week 0) and after the intervention (week 10)
  Concentrations in the brain-derived extracellular vesicles collected from the circulating peripheral blood.

SECONDARY OUTCOMES:
Change in RCAT (Halstead Category Test-Russell Revised Version) | taken at baseline (week 0) and after the intervention (week 10)
  Instrument designed to measure cognitive function. Scores are reported as T-scores while participant's age, gender, ethnicity, and level of education are controlled. A higher T-score correlates to better executive functioning.
Change in Veterans Rand-36 Physical Component Summary (VR-36 PCS) score | taken at baseline (week 0) and after the intervention (week 10)
  Scores reflect physical health-related quality of life. The scores are reported on a scale 0-100 with 0 being the worst possible score and 100 being the best possible score. The mean score of the US population is 50.

CONTACTS AND LOCATIONS:
Overall Officials: Drew A Helmer, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No